CLINICAL TRIAL: NCT04856735
Title: Comparison of the Application of Lidocaine With Intraperitoneal Bupivacaine in Cesarian Operations Wound Infiltration: Randomized, Double-blind, Placebo Controlled Study.
Brief Title: Comparison of the Application of Lidocaine With Intraperitoneal Bupivacaine in Cesarian Operations Wound Infiltration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/384
Record Dates: First submitted 2021-04-14; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Pain; Cesarean Section
MeSH Terms: conditions — Pain, Postoperative | interventions — Cesarean Section; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IPLA:intraperitoneal local anesthetic (Active Comparator): intraperitoneal local anesthetic:after the birth of the newborn and placenta, the uterus is closed and the blood accumulated in the pelvis is carefully wiped with surgical towels, after hemostasis is fully achieved, a total of 20 ml solution containing 10 cc of 0.5% bupivacaine +10 cc 2% lidocaine and 2 injectors containing 20ml saline and the 20ml solution were given to the surgeon. The 20 ml solution containing bupivacaine and lidocaine was injected into the uterine peritoneal region by spraying 5 mL to each quadrant of the uterus before closing the parietal peritoneum or fascia. The parietal peritoneal layer was sutured or left open at the surgeon's preference. At the end of the operation, 20 ml of saline solution was applied subcutaneously in the form of LWI instead of the incision before the skin was closed.
  Interventions: Other: Intraperİtoneal local anaesthesİc İn cesarean sectİon
- LWI:Surgical wound infiltration (Active Comparator): Surgical wound infiltration:a solution containing 20 ml of saline was added to all four quadrants of the uterus in 5 ml volume and 20 ml solution containing lidocaine and bupivacaine were subcutaneously in the form of LWI before the skin was closed.
  Interventions: Other: Local wound infiltrasyon
- C: CONTROL GROUP (Active Comparator): one of the two sterile injectors containing 20 ml of saline was applied to the uterine peritoneal region and the other was applied to the incision area as a local subcutaneous wound infiltration.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Intraperİtoneal local anaesthesİc İn cesarean sectİon — After the birth of the newborn and placenta, the uterus is closed and the blood accumulated in the pelvis is carefully wiped with surgical towels, after hemostasis is fully achieved, a total of 20 ml solution containing 10 cc of 0.5% bupivacaine +10 cc 2% lidocaine and 2 injectors containing 20ml saline and the 20ml solution were given to the surgeon area.
  Other Names: IPLA
  Arms: IPLA:intraperitoneal local anesthetic
Other: Local wound infiltrasyon — A solution containing 20 ml of saline was added to all four quadrants of the uterus in 5 ml volume and 20 ml solution containing lidocaine and bupivacaine were subcutaneously in the form of LWI before the skin was closed
  Other Names: LWI
  Arms: LWI:Surgical wound infiltration
Other: Control group — One of the two sterile injectors containing 20 ml of saline was applied to the uterine peritoneal region and the other was applied to the incision area as a local subcutaneous wound infiltration.
  Other Names: C
  Arms: C: CONTROL GROUP

SUMMARY:
Postoperative pain control is important to reduce morbidity and mortality, and this becomes even more important after cesarean delivery. Severe postpartum pain is associated with chronic pain, and the mother faces a 2.5-fold increased risk of chronic pain and a 3-fold increased risk of postpartum depression compared to mild ones Postoperative pain management is more difficult in the postpartum period. Because the main analgesics used are opioids that are excreted from milk and the newborn may be exposed to the side effects of these drugs . Therefore, multimodal approach is recommended in pain management.

Surgical wound infiltration (LWI) of local anesthetics is an important component of multimodal analgesia . Some of the pain from surgery is caused by an inflammatory response to the surgical incision; therefore, reducing this inflammation can provide a better analgesia and also minimize side effects .

Ease of use and safety of intraperitoneal local anesthetics (IPLA) has been demonstrated in studies and has become a useful alternative to opioid-based analgesic regimens for the treatment of acute postoperative pain.

Investigators aim is to compare the effectiveness of LWI and IPLA applications on postoperative analgesia in women undergoing elective cesarean delivery under spinal anesthesia (SA).

Investigators hypothesis, H0, was that there was no statistically significant difference between the three groups in the mean postoperative pain scores at the 24th hour during movement.

H1 was a statistically significant difference between the mean postoperative pain scores at the 24th hour during the movement between the three groups.

The primary aim of the study was pain scores during the postoperative 24th hour mobilization.

Secondary outcome was total fentanyl consumption (µg) in the first postoperative 24 hours

DETAILED DESCRIPTION:
COMPARISON OF THE APPLICATION OF LIDOCAINE WITH INTRAPERITONEAL BUPIVACAINE IN CESARIAN OPERATIONS WOUND INFILTRATION: RANDOMIZED, DOUBLE-BLIND, PLACEBO CONTROLLED STUDY.

INTRODUCTION The most common surgical procedure in pregnant women is cesarean . Postoperative pain control is important to reduce morbidity and mortality, and this becomes even more important after cesarean delivery. A mother with pain has trouble feeding the newborn . In addition, severe postpartum pain is associated with chronic pain, and the mother faces a 2.5-fold increased risk of chronic pain and a 3-fold increased risk of postpartum depression compared to mild ones .

One of the most important features of a good anesthesia application is a good postoperative pain management. This management is more difficult in the postpartum period. Because the main analgesics used are opioids that are excreted from milk and the newborn may be exposed to the side effects of these drugs . Therefore, multimodal approach is recommended in pain management. In multimodal analgesia, the drugs interact with each other and show a synergistic and additive effect, thus providing better pain control with fewer side effects .

Neuraxial blocks, peripheral nerve blocks, NSAIDS and local anesthetic infiltration of the wound, intraperitoneal local anesthetic delivery were used as part of the multimodal approach.

Surgical wound infiltration (LWI) of local anesthetics is an important component of multimodal analgesia . Some of the pain from surgery is caused by an inflammatory response to the surgical incision; therefore, reducing this inflammation can provide a better analgesia and also minimize side effects .

Ease of use and safety of intraperitoneal local anesthetics (IPLA) has been demonstrated in studies and has become a useful alternative to opioid-based analgesic regimens for the treatment of acute postoperative pain. As an effective adjuvant to postoperative multimodal analgesia, their use in open abdominal operations including gynecological surgery and open abdominal hysterectomy has been reported .

In 1975, Ranney and his friends described intraperitoneal local anesthetic (IPLA) administration in 218 patients who delivered by cesarean section. Although IPLA has received little attention following this publication, recent publications have been shown that IPLA can be used in the treatment of intraoperative pain, prevent postoperative nausea, reduce early postoperative pain and opioid requirements, and shorten hospitalization duration.

Zohar and friends evaluated the effectiveness of IPLA after surgical procedures related to both somatic and visceral pain, and showed that patient-controlled IPLA reduced the need for opioids after bilateral Salpingo-oopherectomy and total abdominal hysterectomy .

Investigators aim is to compare the effectiveness of LWI and IPLA applications on postoperative analgesia in women undergoing elective cesarean delivery under spinal anesthesia (SA).

Investigators hypothesis, H0, was that there was no statistically significant difference between the three groups in the mean postoperative pain scores (VAS scores 0 to 10) at the 24th hour during movement.

H1 was a statistically significant difference between the mean postoperative pain scores at the 24th hour during the movement between the three groups.

The primary aim of the study was pain scores during the postoperative 24th hour mobilization.

Secondary outcome was total fentanyl consumption (µg) in the first postoperative 24 hours.

MATERIALS AND METHODS This prospective randomized placebo-controlled double-blind study was performed on 150 pregnant women aged 18-50 years who underwent a Pfannenstiel incision under spinal anesthesia of ASA I-II, ≥34th gestational week after obtaining the approval of the Atatürk University Medical Faculty Hospital ethics committee and the written consent of patients. to be scheduled. Patients with neuraxial anesthesia contraindications, patients allergic to drugs to be used in the study, BMI> 35 kg / m2, diabetes, preeclampsia, cardiovascular disease, chronic pain and neuropathic pain, patients who have been given opioids in operation due to intraoperative pain, patients with unsuccessful spinal anesthesia who underwent general anesthesia, patients with excessive bleeding during the operation, uterine atony, placement of the drain in the area to be infiltrated, patients who do not want spinal anesthesia, cannot understand VAS, have a history of drug addiction and psychiatric illness will be excluded.

Before the operation, the patients were explained about the procedure, purpose of the study and what VAS was and how it would be used in the postoperative period, and if they feel pain, they could be informed about analgesics at any time after surgery.

After patients have transferred to the operation room, an intravenous (iv) access is obtained with an applicator size of 20 and routine monitorization consisting of electrocardiogram (ECG), peripheral oxygen saturation (SpO2) and non-invasive blood pressure being performed. After the skin is prepared sterile and local infiltration with 2% lidocaine is done, from L3-L4 or L4-L5 range on midline all the patients had received Spinal Anesthesia (SA) and the solution containing 7mg isobaric bupivacaine + 15µg fentanyl was given to the spinal interval in 30 seconds. After the procedure was completed, the patients were placed in the supine position by placing a height under their right hip with a 15 ° left slope. When the sensorial blockade has reached the segments T4-T6 operations were started. All cases were performed with the Pfannenstiel incision. Hypotension was described as systolic blood pressure falling below the basal value by 20%. If hypotension occurs, it will be treated with ephedrine until blood pressure reaches baseline (initial dose 10 mg, intravenously) and rapid colloid or crystalloid infusion. If hypotension persists or recurs, vasopressor treatment will be repeated every 1 minute. Bradycardia will be described as having a heart rate of 50 beats / min and will be treated with 1mg iv atropine.

The patients were randomly assigned equally into Group IPLA, Group LWI and Group C. For this, computerized random numbers table was used. Study drugs were prepared sterile by an anesthesiologist who did not know about the study or did not take part in the evaluation of the study results.

In the group IPLA, after the birth of the newborn and placenta, the uterus is closed and the blood accumulated in the pelvis is carefully wiped with surgical towels, after hemostasis is fully achieved, a total of 20 ml solution containing 10 cc of 0.5% bupivacaine +10 cc 2% lidocaine and 2 injectors containing 20ml saline and the 20ml solution were given to the surgeon. The 20 ml solution containing bupivacaine and lidocaine was injected into the uterine peritoneal region by spraying 5 mL to each quadrant of the uterus before closing the parietal peritoneum or fascia. The parietal peritoneal layer was sutured or left open at the surgeon's preference. At the end of the operation, 20 ml of saline solution was applied subcutaneously in the form of LWI instead of the incision before the skin was closed.

To the group LWI, a solution containing 20 ml of saline was added to all four quadrants of the uterus in 5 ml volume and 20 ml solution containing lidocaine and bupivacaine were subcutaneously in the form of LWI before the skin was closed.

In Group C, one of the two sterile injectors containing 20 ml of saline was applied to the uterine peritoneal region and the other was applied to the incision area as a local subcutaneous wound infiltration.

Study design will be discussed and standardized at a meeting with obstetricians before the start of the research. The study will be blinded because the person administering the study drug did not know which drug was using and the person who evaluated did not know which group was evaluating.

From randomization to completion of statistical analysis, the patient, responsible anesthesiologist and study staff responsible for collecting data will be blinded to the treatment group. The collected data will be stored in a locked cabinet in the anesthesiology department.

Paracetamol 1g and Dexketoprofen 50 mg were administered intravenously to patients 30 minutes before the end of the operation. After the operation, multimodal analgesia was applied to all patients with paracetamol from 15mg / kg every 6 hours for 24 hours and 50 mg dexketoprofen every 12 hours. At the end of the operation, patients started IV PCA. Implemented when 25µg fentanyl iv bolus VAS≥30 was set by adjusting 10 min lock time.

Pain during movement and rest was assessed using the visual analog score (VAS) (0-10).

Nausea and vomiting were evaluated on a scale of 0 to 3. 0 = no nausea or vomiting, 1 = mild nausea that does not require treatment, 2 = moderate nausea that responds to treatment, 3 = severe nausea or vomiting that does not respond to treatment.

Itching was also rated on a scale of 0 to 3. 0 = no itching, 1 = mild itching that does not require treatment, 2 = moderate itching that responds to treatment, and 3 = severe itching that does not respond to treatment.

These evaluations were made at the 2nd, 12th, and 24th hours after intrathecal anesthesia. When nausea and vomiting occurred, 4 mg iv ondansetron was administered and repeated every 8 hours as needed. Pruritus was treated with a 10 mg cetirizine tablet.

Patients' age (years), weight (kg), height (meters), BMI (kg / m2), gestational week, operation time (hour), analgesia duration (hour) (time from spinal anesthesia to the first morphine requirement), cumulative fentanyl consumption (µg) in the first 24 hours postoperatively, number of patients not requiring IV fentanyl, first ambulation time (hour), time of the beginning of bowel movements (hour), local inflammation at the site of the wound, patient satisfaction assessed on a 5-point Likert scale (excellent, very good, good, bad and very bad) 24 hours after surgery were also recorded.

POWER When VAS score is 25 ± 15mm (mean ± std) in the control group and VAS score (mean ± std) is 17 ± 15 (effect size = 0.569) in the study group, the difference between these values can be statistically significant at 80% power and 95% confidence levels in order to be statistically significant, the inclusion of 50 patients in each group was calculated with the G * power program.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* 18-50 years
* ASA I-II,

  -≥34th gestational week
* Exclusion Criteria:
* Patients with neuraxial anesthesia contraindications
* Patients allergic to drugs to be used in the study
* BMI> 35 kg / m2
* Diabetes, preeclampsia, cardiovascular disease, chronic pain and neuropathic pain
* Patients who have been given opioids in operation due to intraoperative pain
* Patients with unsuccessful spinal anesthesia who underwent general anesthesia
* Patients with excessive bleeding during the operation, uterine atony, placement of the drain in the area to be infiltrated
* Patients who do not want spinal anesthesia,
* Cannot understand VAS
* History of drug addiction and psychiatric illness

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant woman
Enrollment: 150 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 24th hours
  The primary outcome in this study is visual analog scores (VAS scores 0 to 10) during mobilization postoperative 24th hour. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
patient satisfaction | 24th hours
  Secondary outcome was total fentanyl consumption (µg) in the first postoperative 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: AYŞENUR DOSTBİL, MD, Study Director — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Betran AP, Merialdi M, Lauer JA, Bing-Shun W, Thomas J, Van Look P, Wagner M. Rates of caesarean section: analysis of global, regional and national estimates. Paediatr Perinat Epidemiol. 2007 Mar;21(2):98-113. doi: 10.1111/j.1365-3016.2007.00786.x. PMID 17302638
- [Background] Klaus MH, Kennell JH, Plumb N, Zuehlke S. Human maternal behavior at the first contact with her young. Pediatrics. 1970 Aug;46(2):187-92. No abstract available. PMID 5432150
- [Background] Nikolajsen L, Sorensen HC, Jensen TS, Kehlet H. Chronic pain following Caesarean section. Acta Anaesthesiol Scand. 2004 Jan;48(1):111-6. doi: 10.1111/j.1399-6576.2004.00271.x. PMID 14674981
- [Background] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Background] Dahl JB, Jeppesen IS, Jorgensen H, Wetterslev J, Moiniche S. Intraoperative and postoperative analgesic efficacy and adverse effects of intrathecal opioids in patients undergoing cesarean section with spinal anesthesia: a qualitative and quantitative systematic review of randomized controlled trials. Anesthesiology. 1999 Dec;91(6):1919-27. doi: 10.1097/00000542-199912000-00045. No abstract available. PMID 10598635